CLINICAL TRIAL: NCT06769126
Title: PRISM: PRecIsion in SCLC Via a Multicohort Study: Randomized Phase II Studies Evaluating Maintenance Durvalumab With or Without Biomarker-Directed Therapy for Extensive Stage Small Cell Lung Cancer (ES-SCLC)
Brief Title: Using Biomarker Tests to Select and Test New, Personalized Treatments for Extensive Stage Small Cell Lung Cancer, PRISM Study
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S2409; NCI-2024-10080 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S2409 (Other: SWOG); S2409 (Other: CTEP); U10CA180888 (NIH)
Record Dates: First submitted 2025-01-02; First posted 2025-01-10 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Extensive Stage Lung Small Cell Carcinoma; Lung Small Cell Carcinoma, A Subtype; Lung Small Cell Carcinoma, I Subtype; Lung Small Cell Carcinoma, N Subtype; Lung Small Cell Carcinoma, P Subtype
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Specimen Handling; ceralasertib; durvalumab; Immunoglobulin G; Disulfides; Etoposide; Magnetic Resonance Spectroscopy; monalizumab; NK Cell Lectin-Like Receptor Subfamily C; Antibodies, Monoclonal, Humanized; Platinum Compounds; AZD5305

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Cohort A, Arm 1 (durvalumab) (Experimental): Patients with ES-SCLC determined to be subtype A or N, and to be SLFN11 positive or patients with subtype P ES-SCLC.
  INDUCTION: Patients may receive a platinum compound plus etoposide per standard care as well as durvalumab IV over 60 minutes on day 1 of each cycle. Cycles repeat every 28 days for 4-6 cycles in the absence of disease progression or unacceptable toxicity.
  CONSOLIDATION: Patients may undergo thoracic radiation as clinically indicated.
  MAINTENANCE: Patients receive durvalumab IV over 60 minutes on day 1 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo CT scan or PET/CT scan and CT scan or MRI throughout the study. Patients also undergo tissue sample collection during screening and may undergo blood sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Biological: Durvalumab; Drug: Etoposide; Procedure: Magnetic Resonance Imaging; Drug: Platinum Compound; Procedure: Positron Emission Tomography; Radiation: Thoracic Radiation Therapy
- Cohort A, Arm 2 (durvalumab, saruparib) (Experimental): Patients with ES-SCLC determined to be subtype A or N, and to be SLFN11 positive or patients with subtype P ES-SCLC.
  INDUCTION: Patients may receive a platinum compound plus etoposide per standard care as well as durvalumab IV over 60 minutes on day 1 of each cycle. Cycles repeat every 28 days for 4-6 cycles in the absence of disease progression or unacceptable toxicity.
  CONSOLIDATION: Patients may undergo thoracic radiation as clinically indicated.
  MAINTENANCE: Patients receive durvalumab IV over 60 minutes on day 1 of each cycle and saruparib PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo CT scan or PET/CT scan and CT scan or MRI throughout the study. Patients also undergo tissue sample collection during screening and may undergo blood sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Biological: Durvalumab; Drug: Etoposide; Procedure: Magnetic Resonance Imaging; Drug: Platinum Compound; Procedure: Positron Emission Tomography; Drug: Saruparib; Radiation: Thoracic Radiation Therapy
- Cohort B, Arm 1 (durvalumab) (Experimental): Patients with ES-SCLC determined to be subtype A or N, and to be SLFN11 negative.
  INDUCTION: Patients may receive a platinum compound plus etoposide per standard care as well as durvalumab IV over 60 minutes on day 1 of each cycle. Cycles repeat every 28 days for 4-6 cycles in the absence of disease progression or unacceptable toxicity.
  CONSOLIDATION: Patients may undergo thoracic radiation as clinically indicated.
  MAINTENANCE: Patients receive durvalumab IV over 60 minutes on day 1 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo CT scan or PET/CT scan and CT scan or MRI throughout the study. Patients also undergo tissue sample collection during screening and may undergo blood sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Biological: Durvalumab; Drug: Etoposide; Procedure: Magnetic Resonance Imaging; Drug: Platinum Compound; Procedure: Positron Emission Tomography; Radiation: Thoracic Radiation Therapy
- Cohort B, Arm 2 (durvalumab, ceralasertib) (Experimental): Patients with ES-SCLC determined to be subtype A or N, and to be SLFN11 negative.
  INDUCTION: Patients may receive a platinum compound plus etoposide per standard care as well as durvalumab IV over 60 minutes on day 1 of each cycle. Cycles repeat every 28 days for 4-6 cycles in the absence of disease progression or unacceptable toxicity.
  CONSOLIDATION: Patients may undergo thoracic radiation as clinically indicated.
  MAINTENANCE: Patients receive durvalumab IV over 60 minutes on day 8 and ceralasertib PO BID on days 1-7 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo CT scan or PET/CT scan and CT scan or MRI throughout the study. Patients also undergo tissue sample collection during screening and may undergo blood sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Drug: Ceralasertib; Procedure: Computed Tomography; Biological: Durvalumab; Drug: Etoposide; Procedure: Magnetic Resonance Imaging; Drug: Platinum Compound; Procedure: Positron Emission Tomography; Radiation: Thoracic Radiation Therapy
- Cohort C, Arm 1 (durvalumab) (Experimental): Patients with ES-SCLC determined to be subtype I.
  INDUCTION: Patients may receive a platinum compound plus etoposide per standard care as well as durvalumab IV over 60 minutes on day 1 of each cycle. Cycles repeat every 28 days for 4-6 cycles in the absence of disease progression or unacceptable toxicity.
  CONSOLIDATION: Patients may undergo thoracic radiation as clinically indicated.
  MAINTENANCE: Patients receive durvalumab IV over 60 minutes on day 1 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo CT scan or PET/CT scan and CT scan or MRI throughout the study. Patients also undergo tissue sample collection during screening and may undergo blood sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Biological: Durvalumab; Drug: Etoposide; Procedure: Magnetic Resonance Imaging; Drug: Platinum Compound; Procedure: Positron Emission Tomography; Radiation: Thoracic Radiation Therapy
- Cohort C, Arm 2 (durvalumab, monalizumab) (Experimental): Patients with ES-SCLC determined to be subtype I.
  INDUCTION: Patients may receive a platinum compound plus etoposide per standard care as well as durvalumab IV over 60 minutes on day 1 of each cycle. Cycles repeat every 28 days for 4-6 cycles in the absence of disease progression or unacceptable toxicity.
  CONSOLIDATION: Patients may undergo thoracic radiation as clinically indicated.
  MAINTENANCE: Patients receive durvalumab IV over 60 minutes on day 1 and monalizumab IV over 60 minutes on days 1 and 15 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo CT scan or PET/CT scan and CT scan or MRI throughout the study. Patients also undergo tissue sample collection during screening and may undergo blood sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Biological: Durvalumab; Drug: Etoposide; Procedure: Magnetic Resonance Imaging; Biological: Monalizumab; Drug: Platinum Compound; Procedure: Positron Emission Tomography; Radiation: Thoracic Radiation Therapy

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo tissue and blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Ceralasertib — Given PO
  Other Names: AZD6738
  Arms: Cohort B, Arm 2 (durvalumab, ceralasertib)
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Biological: Durvalumab — Given IV
  Other Names: Imfinzi; Immunoglobulin G1, Anti-(Human Protein B7-H1) (Human Monoclonal MEDI4736 Heavy Chain), Disulfide with Human Monoclonal MEDI4736 Kappa-chain, Dimer; MEDI 4736; MEDI-4736; MEDI4736
Drug: Etoposide — Given etoposide
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16; VP 16-213; VP 16213; VP-16; VP-16-213; VP-16213; VP16; VP16213
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Biological: Monalizumab — Given IV
  Other Names: Immunoglobulin G4-kappa, Anti-(Homo sapiens KLRC1 (Killer Cell Lectin-like Receptor Subfamily C Member 1, NKG2-a, NKG2a, CD159A, CD94)), Humanized Monoclonal Antibody; IPH-2201; IPH2201; NN-8765; NN8765; NN8765-3658
  Arms: Cohort C, Arm 2 (durvalumab, monalizumab)
Drug: Platinum Compound — Given platinum compound
  Other Names: Platinum Agents; Platinum-Based Chemotherapeutic Agent
Procedure: Positron Emission Tomography — Undergo PET/CT scan
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT
Drug: Saruparib — Given PO
  Other Names: AZD 5305; AZD-5305; AZD5305; PARP Inhibitor AZD5305
  Arms: Cohort A, Arm 2 (durvalumab, saruparib)
Radiation: Thoracic Radiation Therapy — Undergo thoracic radiation
  Other Names: Thoracic Radiotherapy

SUMMARY:
This phase II trial tests how well biomarker tests on patients tumor tissue works in selecting personalized treatments for patients with extensive stage small cell lung cancer (ES-SCLC). Biomarker tests look for certain features in cancer cells that may give doctors more information about what is driving cancer and how to treat it. Based on the biomarker test results, study doctors can determine the subtype of ES-SCLC that study treatments can target. This study also tests different types of maintenance treatment for ES-SCLC with drugs durvalumab, saruparib, ceralasertib or monalizumab. Maintenance treatment is given after initial treatment and is given to help keep the cancer under control and prevent it from getting worse. Immunotherapy with monoclonal antibodies, such as durvalumab and monalizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Saruparib is a PARP inhibitor. PARP is a protein that helps repair damaged deoxyribonucleic acid (DNA). Blocking PARP may prevent cancer cells from repairing their damaged DNA, causing them to die. PARP inhibitors are a type of targeted therapy. Ceralasertib may stop the growth of tumor cells and may kill them by blocking some of the enzymes needed for tumor cell growth. Giving biomarker selected personalized maintenance treatment with durvalumab, saruparib, ceralasertib or monalizumab may work better in treating patients with ES-SCLC.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To test participants' tissue specimens to determine their eligibility to 1 of the 3 treatment cohorts created based on their small cell lung cancer (SCLC) subtype and SLFN11 status. (Screening) II. To compare progression-free survival (PFS) in participants with extensive stage SCLC (ES-SCLC) (subtypes A or N & SLFN11 positive) or ES-SCLC (subtype P) randomized to durvalumab (MEDI4736) with or without saruparib (AZD5305) as maintenance therapy following induction chemoimmunotherapy with platinum, etoposide, and durvalumab (MEDI4736). (Cohort A) III. To compare PFS in participants with ES-SCLC subtypes A or N & SLFN11 negative randomized to durvalumab with or without ceralasertib (AZD6738) as maintenance therapy following induction chemoimmunotherapy with cisplatin or carboplatin, etoposide, and durvalumab (MEDI4736). (Cohort B) IV. To compare PFS participants with ES-SCLC subtype I randomized to durvalumab (MEDI4736) with or without monalizumab (IPH2201) as maintenance therapy following induction chemoimmunotherapy with cisplatin or carboplatin, etoposide, and durvalumab (MEDI4736). (Cohort C)

SECONDARY OBJECTIVES:

I. To evaluate the percentage of participant tissue that are able to have SCLC subtype status determined. (Screening) II. To evaluate the percentage of participant tissue that are able to have SLFN11 status determined. (Screening) III. To estimate the percentage of participants assigned to a cohort that register to be randomized. (Screening) IV. To evaluate the safety of saruparib (AZD5305) in combination with durvalumab by estimating the rate of dose limiting toxicities reported during the first cycle of treatment in the safety-run-in population. (Cohort A) V. To compare PFS between the arms in the subset of participants with A or N subtype and SLFN11 positive. (Cohort A) VI. To compare overall survival (OS) between the arms. (Cohort A) VII. To evaluate the frequency and severity of toxicities by Common Terminology Criteria for Adverse Events (CTCAE) within each treatment arm. (Cohort A) VIII. To compare OS between the arms. (Cohort B) IX. To evaluate the frequency and severity of toxicities by CTCAE within each arm. (Cohort B) X. To compare OS between the arms. (Cohort C) XI. To evaluate the frequency and severity of toxicities by CTCAE within each arm. (Cohort C)

TRANSLATIONAL MEDICINE OBJECTIVE:

I. To bank specimens for future correlative studies.

OUTLINE:

INDUCTION: Patients may receive a platinum compound plus etoposide per standard care as well as durvalumab intravenously (IV) over 60 minutes on day 1 of each cycle. Cycles repeat every 28 days for 4-6 cycles in the absence of disease progression or unacceptable toxicity.

CONSOLIDATION: Patients may undergo thoracic radiation as clinically indicated.

MAINTENANCE: Patients are assigned to 1 of 3 cohorts and then randomized to 1 of 2 arms within each cohort to which they were assigned.

COHORT A: Patients with ES-SCLC determined to be subtype A or N, and to be SLFN11 positive or patients with subtype P ES-SCLC.

ARM 1: Patients receive durvalumab IV over 60 minutes on day 1 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARM 2: Patients receive durvalumab IV over 60 minutes on day 1 of each cycle and saruparib orally (PO) once daily (QD) on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

COHORT B: Patients with ES-SCLC determined to be subtype A or N, and to be SLFN11 negative.

ARM 1: Patients receive durvalumab IV over 60 minutes on day 1 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARM 2: Patients receive durvalumab IV over 60 minutes on day 8 and ceralasertib PO twice daily (BID) on days 1-7 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

COHORT C: Patients with ES-SCLC determined to be subtype I.

ARM 1: Patients receive durvalumab IV over 60 minutes on day 1 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARM 2: Patients receive durvalumab IV over 60 minutes on day 1 and monalizumab IV over 60 minutes on days 1 and 15 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Additionally, patients undergo computed tomography (CT) scan or positron emission tomography (PET)/CT scan and CT scan or magnetic resonance imaging (MRI) throughout the study. Patients also undergo tissue sample collection during screening and may undergo blood sample collection throughout the study.

After completion of study treatment, patients are followed up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* STEP 1: SCREENING AND INDUCTION TREATMENT REGISTRATION: Participants must not have a prior or concurrent malignancy whose natural history or treatment (in the opinion of the treating physician) has the potential to interfere with the safety or efficacy assessment of the investigational regimen
* STEP 1: SCREENING AND INDUCTION TREATMENT REGISTRATION: Participants must not have a history of limited stage small cell lung cancer
* STEP 1: SCREENING AND INDUCTION TREATMENT REGISTRATION: Participants must meet 1 of the following criteria prior to step 1:

  * Treatment naïve and planning to receive frontline induction treatment with platinum plus etoposide in combination with durvalumab, OR,
  * Have initiated frontline induction therapy and completed at least 1 (≥ 1) cycle and at most 3 (≤ 3) cycles of platinum and etoposide. At most 2 (≤ 2) of these cycles could have been given without durvalumab

    * NOTE: Participants must not have received immunotherapy other than durvalumab (e.g., atezolizumab) prior to enrollment
* STEP 1: SCREENING AND INDUCTION TREATMENT REGISTRATION: Participants must not have received any anti PD-1 or anti PD-L1 (including durvalumab [MEDI4736]) treatment for SCLC prior to starting frontline induction treatment for ES-SCLC
* STEP 1: SCREENING AND INDUCTION TREATMENT REGISTRATION: Participants must not have received anti PD-1 or anti PD-L1 other than durvalumab (MEDI4736) as part of frontline induction treatment for ES-SCLC. Participants must have not received atezolizumab, pembrolizumab, or nivolumab as part of frontline induction treatment
* STEP 1: SCREENING AND INDUCTION TREATMENT REGISTRATION: Participants must not have received any investigational agent for the treatment of ES-SCLC
* STEP 1: SCREENING AND INDUCTION TREATMENT REGISTRATION: Participants must not be planning to receive any concurrent non-protocol directed chemotherapy, immunotherapy, biologic or hormonal therapy for SCLC treatment while receiving treatment on this study

  * NOTE: If participant has bone metastases, bisphosphonates are allowed
* STEP 1: SCREENING AND INDUCTION TREATMENT REGISTRATION: Participants must not have any unresolved toxicity National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) grade ≥ 2 from previous anticancer therapy with the exception of alopecia, and vitiligo
* STEP 1: SCREENING AND INDUCTION TREATMENT REGISTRATION: Participants must be ≥ 18 years old at the time of step 1 registration
* STEP 1: SCREENING AND INDUCTION TREATMENT REGISTRATION: Participants must be able to safely receive the frontline induction treatment with platinum plus etoposide in combination with durvalumab, per the current Food and Drug Administration (FDA)-approved package insert(s), institutional guidelines, and the treating investigator's discretion
* STEP 1: SCREENING AND INDUCTION TREATMENT REGISTRATION: Participants must have Zubrod performance status of 0-2 within 28 days prior to step 1 registration
* STEP 1: SCREENING AND INDUCTION TREATMENT REGISTRATION: Participants must have fully recovered from the effects of prior surgery in the opinion of the treating investigator within 28 days prior to step 1 registration
* STEP 1: SCREENING AND INDUCTION TREATMENT REGISTRATION: Participants must not have had an allogenic organ transplantation
* STEP 1: SCREENING AND INDUCTION TREATMENT REGISTRATION: Participants must not have medical contraindications to receiving immunotherapy, including history of non-infectious pneumonitis that required steroids or active autoimmune disease that has required systemic treatment with disease modifying agents, corticosteroids or immunosuppressive drugs in the past two years. Replacement therapy (e.g. thyroxine for pre-existing hypothyroidism, insulin for type I diabetes mellitus, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment. Intra-articular steroid injections are allowed
* STEP 1: SCREENING AND INDUCTION TREATMENT REGISTRATION: Participants must not be pregnant or nursing (nursing includes breast milk fed to an infant by any means, including from the breast, milk expressed by hand, or pumped). Individuals who are of reproductive potential must have agreed to use an effective contraceptive method during protocol therapy and for 6 months following completion of protocol therapy with details provided as a part of the consent process. A person who has had menses at any time in the preceding 12 consecutive months or who has semen likely to contain sperm is considered to be of "reproductive potential." In addition to routine contraceptive methods, "effective contraception" also includes refraining from sexual activity that might result in pregnancy and surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention) including hysterectomy, bilateral oophorectomy, bilateral tubal ligation/occlusion, and vasectomy with testing showing no sperm in the semen. Participants should not breastfeed during protocol therapy and for 6 months following completion of protocol therapy
* STEP 1: SCREENING AND INDUCTION TREATMENT REGISTRATION: Participants must have adequate tumor tissue available from SCLC and agree to have these tissue specimens submitted. Participants must agree to have any leftover tissue (tissue that remains after subtype and biomarker testing) retained for the use of future correlative studies.

  * NOTE: After a participant has been registered to step 1 registration, the tissue must be submitted to BostonGene. Sites will receive a notification from the Southwest Oncology Group (SWOG) Statistics and Data Management Center within 19 days after tissue submission. Patients must not be registered to step 2 prior to receiving notification of cohort assignment
  * NOTE: A histologic review will be performed to confirm adequate cellularity for the testing. If inadequate cellularity, additional archival unstained slides from the same participant may be submitted if it does not exceed the window of starting maintenance therapy
* STEP 1: SCREENING AND INDUCTION TREATMENT REGISTRATION: NOTE: As a part of the Oncology Patient Enrollment Network (OPEN) registration process the treating institution's identity is provided in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered in the system.

  * Participants must be informed of the investigational nature of this study and must sign and give informed consent in accordance with institutional and federal guidelines. For participants with impaired decision-making capabilities, legally authorized representatives may sign and give informed consent on behalf of study participants in accordance with applicable federal, local, and Central Institutional Review Board (CIRB) regulations
* STEP 2: COHORT REGISTRATION AND MAINTENANCE RANDOMIZATION: Site must have received notification from the SWOG Statistics and Data Management Center (SDMC) of the participant's SLFN11 testing results and have been determined to have subtype A, N, I, or P: confirmed by BostonGene and assigned to a cohort
* STEP 2: COHORT REGISTRATION AND MAINTENANCE RANDOMIZATION: Participants may have measurable or non-measurable disease per Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1) and must have their disease assessed by CT of chest/abdomen/pelvis (with contrast unless contraindicated) within 28 days prior to step 2 for measurable disease or within 42 days prior to step 2 for non-measurable disease. All known sites of disease must be assessed and documented on the baseline tumor assessment form (RECIST 1.1). Any lesions assessed using a non-diagnostic PET/CT of chest/abdomen/pelvis will be considered non-measurable lesions
* STEP 2: COHORT REGISTRATION AND MAINTENANCE RANDOMIZATION: Participants must have a CT or MRI scan of the brain to evaluate for central nervous system (CNS) disease within 42 days prior to step 2 randomization. Participant must not have leptomeningeal disease, spinal cord compression, or symptomatic brain metastases unless: (1) metastases have been locally treated and have remained clinically controlled and asymptomatic for at least 14 days following treatment, and prior to step 2 randomization, AND (2) participant has no residual neurological dysfunction and has been off corticosteroids for at least 24 hours prior to step 2 randomization
* STEP 2: COHORT REGISTRATION AND MAINTENANCE RANDOMIZATION: Participants with untreated brain metastases must be asymptomatic and stable off steroids prior to step 2 randomization.

  * NOTE: Exceptions to corticosteroid criterion are: (1) intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra-articular injection), (2) systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent, or (3) steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication). Premedication with steroids for chemotherapy is acceptable
* STEP 2: COHORT REGISTRATION AND MAINTENANCE RANDOMIZATION: Participants must not have experienced disease progression in the opinion of treating investigator during induction treatment and prior to step 2
* STEP 2: COHORT REGISTRATION AND MAINTENANCE RANDOMIZATION: Participants must have completed frontline induction therapy. Induction therapy must have included 4-6 cycles of platinum plus etoposide and 4 cycles of durvalumab (MEDI4736); at most 2 (≤ 2) cycles of platinum plus etoposide may have been given without durvalumab (MEDI4736). Durvalumab (MEDI4736) must have been given in combination with platinum plus etoposide
* STEP 2: COHORT REGISTRATION AND MAINTENANCE RANDOMIZATION: Participants who received consolidation thoracic radiation therapy must have completed all radiation therapy at least 14 days prior to step 2
* STEP 2: COHORT REGISTRATION AND MAINTENANCE RANDOMIZATION: For participants not receiving consolidation thoracic radiation, step 2 registration must occur at least 3 weeks but not more than 6 weeks after the last dose of frontline induction therapy (platinum plus etoposide in combination with durvalumab [MEDI4736])
* STEP 2: COHORT REGISTRATION AND MAINTENANCE RANDOMIZATION: For participants receiving consolidation thoracic radiation after induction therapy, step 2 registration must occur at least 3 weeks but no more than 8 weeks after the last dose of frontline induction therapy (platinum plus etoposide in combination with durvalumab [MEDI4736])
* STEP 2: COHORT REGISTRATION AND MAINTENANCE RANDOMIZATION: Participants must not have received atezolizumab, pembrolizumab, or nivolumab as part of their frontline induction treatment. Participants must not have received prophylactic cranial irradiation (PCI)
* STEP 2: COHORT REGISTRATION AND MAINTENANCE RANDOMIZATION: Participants must have a complete medical history and physical within 28 days prior to step 2
* STEP 2: COHORT REGISTRATION AND MAINTENANCE RANDOMIZATION: Participants must have body weight > 30 kg
* STEP 2: COHORT REGISTRATION AND MAINTENANCE RANDOMIZATION: Participants must have Zubrod performance status of 0-2 within 28 days prior to step 2
* STEP 2: COHORT REGISTRATION AND MAINTENANCE RANDOMIZATION: Hemoglobin > 9.0 g/dL (within 28 days prior to step 2)
* STEP 2: COHORT REGISTRATION AND MAINTENANCE RANDOMIZATION: Absolute neutrophil count ≥ 1.5 x 10^3/uL (within 28 days prior to step 2)
* STEP 2: COHORT REGISTRATION AND MAINTENANCE RANDOMIZATION: Platelets ≥ 100 x 10^3/uL (within 28 days prior to step 2)
* STEP 2: COHORT REGISTRATION AND MAINTENANCE RANDOMIZATION: Total bilirubin ≤ institutional upper limit of normal (ULN) unless history of Gilbert's disease. Participants with history of Gilbert's disease must have total bilirubin ≤ 5 x institutional ULN (within 28 days prior to step 2)
* STEP 2: COHORT REGISTRATION AND MAINTENANCE RANDOMIZATION: Aspartate aminotransferase (AST)/alanine transaminase (ALT) ≤ 5 × institutional ULN (within 28 days prior to step 2)
* STEP 2: COHORT REGISTRATION AND MAINTENANCE RANDOMIZATION: Participants must have creatinine ≤ 1.5x the institutional upper limit of normal (IULN) OR measured OR calculated creatinine clearance ≥ 45 mL/min using the following Cockcroft-Gault Formula For creatinine clearance formula see the tools on the Cancer Research and Biostatistics (CRA) Workbench https://txwb.crab.org/TXWB/Tools.aspx
* STEP 2: COHORT REGISTRATION AND MAINTENANCE RANDOMIZATION: Participants with a known history of human immunodeficiency virus (HIV)-infection must be on effective anti-retroviral therapy at registration and have undetectable viral load test on the most recent test results obtained within 6 months prior to step 2 registration
* STEP 2: COHORT REGISTRATION AND MAINTENANCE RANDOMIZATION: Participants with a known history of chronic hepatitis B virus (HBV) infection must have undetectable HBV viral load while on suppressive therapy on the most recent test results obtained within 6 months prior to randomization, if indicated
* STEP 2: COHORT REGISTRATION AND MAINTENANCE RANDOMIZATION: Participants with a known history of hepatitis C virus (HCV) infection must have been treated and cured or currently be receiving treatment for HVC. Participants currently being treated for HCV infection must have undetectable HCV viral load test on the most recent test results obtained within 6 months prior to randomization, if indicated
* STEP 2: COHORT REGISTRATION AND MAINTENANCE RANDOMIZATION: Participants must not have experienced the following during induction treatment: Any grade 3 or worse immune-mediated adverse event (irAE) (except asymptomatic nonbullous/nonexfoliative rash) or any unresolved grade 2 irAE, nor have experienced a toxicity that led to permanent discontinuation of prior durvalumab (MEDI4736). Toxicity of any grade that requires replacement therapy and has stabilized on therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is allowed
* STEP 2: COHORT REGISTRATION AND MAINTENANCE RANDOMIZATION: Participants must not be pregnant or nursing (nursing includes breast milk fed to an infant by any means, including from the breast, milk expressed by hand, or pumped). Individuals who are of reproductive potential must have agreed to use an effective contraceptive method during protocol therapy and for 6 months following completion of protocol therapy with details provided as a part of the consent process. A person who has had menses at any time in the preceding 12 consecutive months or who has semen likely to contain sperm is considered to be of "reproductive potential." In addition to routine contraceptive methods, "effective contraception" also includes refraining from sexual activity that might result in pregnancy and surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention) including hysterectomy, bilateral oophorectomy, bilateral tubal ligation/occlusion, and vasectomy with testing showing no sperm in the semen. Participants should not breastfeed during protocol therapy and for 6 months following completion of protocol therapy
* STEP 2: COHORT REGISTRATION AND MAINTENANCE RANDOMIZATION: Participants must not have received a live or live attenuated vaccine within 30 days prior to step 2. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster, yellow fever rabies, Bacillus Calmette-Guerin (BCG) and typhoid vaccine. Seasonal influenza vaccines and COVID-19 vaccines are allowed, however, intranasal influenza vaccines (e.g. Flu-Mist) are live attenuated, and are not allowed
* STEP 2: COHORT REGISTRATION AND MAINTENANCE RANDOMIZATION: Participants must be offered the opportunity to participate in specimen banking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2025-11-06 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Screen success rate (Screening) | Up to 3 years
  Will test participants' tissue specimens to determine their eligibility to 1 of the 3 treatment cohorts created based on their small cell lung cancer (SCLC) subtype and SLFN11 status. Will evaluate rate of participants who successfully get a cohort assignment based on SCLC subtype and SLNFN11 status, as appropriate.
Progression-free survival (PFS) (Cohort A) | From date of randomization to treatment within a cohort to date of first documentation of progression, symptomatic deterioration, or death due to any cause, assessed up to 3 years
  Will compare PFS in participants with extensive stage SCLC (ES-SCLC) (subtypes A or N & SLFN11 positive) or ES-SCLC (subtype P) randomized to durvalumab (MEDI4736) with or without saruparib (AZD5305) as maintenance therapy following induction chemoimmunotherapy with platinum, etoposide, and durvalumab (MEDI4736). Will be estimated using the Kaplan-Meier method. Associated confidence intervals about the median will be performed using the Brookmeyer-Crowley method. Binary proportions and associated confidence intervals will be calculated.
PFS (Cohort B) | From date of randomization to treatment within a cohort to date of first documentation of progression, symptomatic deterioration, or death due to any cause, assessed up to 3 years
  Will compare PFS in participants with ES-SCLC subtypes A or N and SLFN11 negative randomized to durvalumab with or without ceralasertib (AZD6738) as maintenance therapy following induction chemoimmunotherapy with cisplatin or carboplatin, etoposide, and durvalumab (MEDI4736). Will be estimated using the Kaplan-Meier method. Associated confidence intervals about the median will be performed using the Brookmeyer-Crowley method.
PFS (Cohort C) | From date of randomization to treatment within a cohort to date of first documentation of progression, symptomatic deterioration, or death due to any cause, assessed up to 3 years
  Will compare PFS participants with ES-SCLC subtype I randomized to durvalumab (MEDI4736) with or without monalizumab (IPH2201) as maintenance therapy following induction chemoimmunotherapy with cisplatin or carboplatin, etoposide, and durvalumab (MEDI4736). Will be estimated using the Kaplan-Meier method. Associated confidence intervals about the median will be performed using the Brookmeyer-Crowley method.

SECONDARY OUTCOMES:
SCLC subtype status (Screening) | Up to 3 years
  Will evaluate the percentage of participant tissue that are able to have SCLC subtype status determined.
SLFN11 status (Screening) | Up to 3 years
  Will evaluate the percentage of participant tissue that are able to have SLFN11 status determined.
Assigned to a cohort and register to be randomized (Screening) | Up to 3 years
  Will estimate the percentage of participants assigned to a cohort that register to be randomized.
Incidence of dose limiting toxicity (DLT) (Cohort A, safety run-in) | During the first cycle of treatment (each cycle is 28 days)
  Will evaluate the safety of saruparib (AZD5305) in combination with durvalumab by estimating the rate of DLTs in the safety-run-in population. Will be assessed by treatment-related grade 3 or higher non hematologic toxicity, treatment-related grade 4 or higher hematologic toxicity, or any grade of treatment-related toxicity that in the opinion of the treating physician directly leads to that participant decision to drug discontinuation.
PFS (Cohort A) | From date of randomization to treatment within a cohort to date of first documentation of progression, symptomatic deterioration, or death due to any cause, assessed up to 3 years
  Will compare PFS between the arms in the subset of participants with A or N subtype and SLFN11 positive. Will be estimated using the Kaplan-Meier method. Associated confidence intervals about the median will be performed using the Brookmeyer-Crowley method. Binary proportions and associated confidence intervals will be calculated.
Overall survival (OS) (Cohort A) | From date of randomization to treatment within a cohort to date of death due to any cause, assessed up to 3 years
  Will compare OS between the arms. Will be estimated using the Kaplan-Meier method. Associated confidence intervals about the median will be performed using the Brookmeyer-Crowley method. Binary proportions and associated confidence intervals will be calculated.
Incidence of adverse events (Cohort A) | Up to 3 years
  Will evaluate the frequency and severity of toxicities by Common Terminology Criteria for Adverse Events(CTCAE) within each treatment arm.
OS (Cohort B) | From date of randomization to treatment within a cohort to date of death due to any cause, assessed up to 3 years
  Will compare OS between the arms. Will be estimated using the Kaplan-Meier method. Associated confidence intervals about the median will be performed using the Brookmeyer-Crowley method.
Incidence of adverse events (Cohort B) | Up to 3 years
  Will evaluate the frequency and severity of toxicities by CTCAE within each arm.
OS (Cohort C) | From date of randomization to treatment within a cohort to date of death due to any cause, assessed up to 3 years
  Will compare OS between the arms. Will be estimated using the Kaplan-Meier method. Associated confidence intervals about the median will be performed using the Brookmeyer-Crowley method.
Incidence of adverse events (Cohort C) | Up to 3 years
  Will evaluate the frequency and severity of toxicities by CTCAE within each arm.

OTHER OUTCOMES:
Bank specimens | Up to 3 years
  Will bank specimens for future correlative studies.

CONTACTS AND LOCATIONS:
Overall Officials: Anne C Chiang, Principal Investigator — SWOG Cancer Research Network
Locations (50):
- United States (50):
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Loyola University Medical Center, Maywood, Illinois
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - UI Health Care Mission Cancer and Blood - Ankeny Clinic, Ankeny, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - McFarland Clinic - Trinity Cancer Center, Fort Dodge, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - UI Health Care Mission Cancer and Blood - Waukee Clinic, Waukee, Iowa
  - The Iowa Clinic PC, West Des Moines, Iowa
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Community Medical Center, Missoula, Montana
  - FirstHealth of the Carolinas-Moore Regional Hospital, Pinehurst, North Carolina
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Duluth Clinic Ashland, Ashland, Wisconsin